CLINICAL TRIAL: NCT01037062
Title: An Open-Label Rollover Study of Entecavir (BMS-200475) in Adults With Chronic Hepatitis B Infection Who Have Completed Previous Phase II Studies in Japan But Who Require Further Treatment
Brief Title: An Open-Label Rollover Study of Entecavir (BMS-200475) in Adults With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-060
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Entecavir (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablet, P.O. 0.5, 1 mg, once daily
  Other Names: Baraclude; BMS-200475

SUMMARY:
To provide open-label entecavir to subjects who have completed previous blinded entecavir trials in Japan and are assessed by the investigator as likely to benefit from additional anti-hepatitis B therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed a previous entecavir Phase II studies (AI463047, 052 or 053);
* ALT ≤ 10 x upper limit of normal;
* Subjects must have well-compensated liver disease according to ALL of the following criteria;

  1. Prothrombin time ≤ 3 seconds prolonged compared to control value or INR ≤ 1.5
  2. Serum albumin ≥ 3 g/dL (≥ 30 g/L)
  3. Serum bilirubin ≤ 2.5 mg/dL (≤ 42.75 μmol/L)

Exclusion Criteria:

* Sex and Reproductive Status Exceptions
* Target Disease Exceptions
* Medical History and Concurrent Diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To provide open-label entecavir to subjects who have completed previous blinded entecavir trials in Japan and are assessed by the investigator as likely to benefit from additional anti-hepatitis B therapy | 24 weeks

SECONDARY OUTCOMES:
Incidence of clinical adverse events and discontinuations due to adverse events of entecavir for each cohort | Week 2, 4, 6, 8, 10, 12, 16, 20 and 24 post dosing
Incidence of laboratory abnormalities of of entecavir for each cohort | Week 2, 4, 6, 8, 10, 12, 16, 20 and 24 post dosing
Proportion of subjects HBeAg-positive at baseline who have loss of HBeAg from serum | Day 1, Week 12, Week 24 and every subsequent 24 week during dosing
Proportion of subjects HBeAg-positive at baseline who achieve seroconversion (loss of HBeAg and appearance of HBeAb) | Day 1, Week 12, Week 24 and every subsequent 24 week during dosing
Proportion of subjects with abnormal ALT at baseline who achieve normalization of serum ALT at Week 48 | Day 1, Week 48
Proportion of subjects who achieve HBV DNA levels by PCR assay less than the limit of quantification (LOQ) | Day 1, Week 12, 24, and subsequent 24 week during dosing
Proportion of subjects positive for HBeAg at baseline who achieve HBV DNA levels by PCR assay less than LOQ, normal serum ALT, and seroconversion | Week 8, 16, 24 post dosing
Proportion of subjects negative for HBeAg at baseline who achieve HBV DNA levels by PCR assay less than LOQ and normal ALT and remain negative for HBeAg | Day 1, Week 12, Week 24 and every subsequent 24 weeks during dosing
Proportion of subjects who achieved Complete Response during therapy, who have sustained Complete Response for 24 weeks after stopping drug | 24 Week post dosing
Proportion of subjects with histological improvement in the liver at Wks 48 & 96 [improvement in necroinflammatory score and no worsening of fibrosis at Wks 48 & 96 liver biopsy compared to baseline & to baseline in previous study] | Week 48, 96
NChanges in liver histology as assessed by the New Inuyama Classification for histological assessment of chronic hepatitis | Week 48 & Week 96
Incidence of genotypic changes in HBV DNA polymerase conferring resistance to entecavir in subjects with confirmed ≥1 log10 increase in HBV DNA from nadir on treatment | Week 2, 4, ± days, Week 8 every 4 weeks ± 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- Japan (39):
  - Local Institution, Aichi-Gun, Aichi-ken
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Onsen-Gun, Ehime
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Gifu, Gifu
  - Local Institution, Ogaki-Shi, Gifu
  - Local Institution, Fukuyama-Shi, Hiroshima
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Asahikawa-Shi, Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Akashi-Shi, Hyōgo
  - Local Institution, Morioka, Iwate
  - Local Institution, Mitoyo-Gun, Kagawa-ken
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Miyazaki-Gun, Miyazaki
  - Local Institution, Matsumoto, Nagano
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Omura-Shi, Nagasaki
  - Local Institution, Niigata, Niigata
  - Local Institution, Oita-Gun, Oita Prefecture
  - Local Institution, Kurashiki-Shi, Okayama-ken
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Tsuyama-Shi, Okayama-ken
  - Local Institution, Kawachinagano-Shi, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Sakai-Shi, Osaka
  - Local Institution, Suita-Shi, Osaka
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Minato-Ku, Tokyo
  - Local Institution, Musashino-Shi, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Tokyo, Tokyo
  - Local Institution, Ube-Shi, Yamaguchi
  - Local Institution, Nakakoma-Gun, Yamanashi

REFERENCES:
- [Background] Yokosuka O, Takaguchi K, Fujioka S, Shindo M, Chayama K, Kobashi H, Hayashi N, Sato C, Kiyosawa K, Tanikawa K, Ishikawa H, Masaki N, Seriu T, Omata M. Long-term use of entecavir in nucleoside-naive Japanese patients with chronic hepatitis B infection. J Hepatol. 2010 Jun;52(6):791-9. doi: 10.1016/j.jhep.2009.12.036. Epub 2010 Mar 24. PMID 20409606
- [Background] Karino Y, Toyota J, Kumada H, Katano Y, Izumi N, Kobashi H, Sata M, Moriyama M, Imazeki F, Kage M, Ishikawa H, Masaki N, Seriu T, Omata M. Efficacy and resistance of entecavir following 3 years of treatment of Japanese patients with lamivudine-refractory chronic hepatitis B. Hepatol Int. 2010 Feb 6;4(1):414-22. doi: 10.1007/s12072-009-9162-x. PMID 20305760
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx